CLINICAL TRIAL: NCT06177132
Title: Vestibular Infant Screening - Rehabilitation (VIS-REHAB): Protocol for a Randomised Controlled Trial on Vestibular Rehabilitation Therapy (VRT) in Vestibular-impaired Children
Brief Title: Vestibular Infant Screening - Rehabilitation
Acronym: VIS-REHAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIS-REHAB
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vestibular Disorder
Keywords: Therapy; Vestibular Rehabilitation Therapy; VRT; Gaze stability; Postural control
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Two-parallel group, superiority, randomised controlled crossover trial with 1:1 allocation ratio
Who Masked: Outcomes Assessor
Masking Description: Participants cannot be blinded to their assigned groups, as they will be aware of the protocol received at any given time. The assessment of primary and secondary outcome measures will be conducted by a separate outcome assessor who will be blinded to patient allocation. Data analysis procedures will not involve blinding since they will be performed by the same individual responsible for conducting the rehabilitation sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VIS-REHAB Protocol (Experimental): The VIS-REHAB protocol entails 30-minute sessions conducted twice a week over a span of 9 weeks. These sessions are structured with 20 minutes dedicated to enhancing postural stability and 10 minutes focused on improving gaze stability. In greater detail, a minimum of 5 minutes time is reserved for counselling and providing background information on the exercises, focused on the vestibular issue. Apart from the counselling part, each session consist of 3 different exercise categories ((static postural stability, dynamic postural stability, general gross motor training (focus on PS), oculomotor function, gaze stability, or general gross motor training (focus on GS)), each carried out for 5 to 10 minutes.
  Interventions: Behavioral: VIS-REHAB protocol
- CTRL Protocol (No Intervention): In the control (CTRL) protocol, all forms of physical therapy in the context of motor development are ceased. Occupational therapy, speech-language therapy and physical therapy for other purposes are not covered by this commitment. Additionally, the child and parents are asked to not do any home exercises on their own. However, sports activities and other recreational hobbies will not be asked to be temporary halted, since they will be continued in the active rehabilitation programme as well.

INTERVENTIONS:
Behavioral: VIS-REHAB protocol — The VIS-REHAB protocol entails two essential components: postural stability (PS) and gaze stability (GS). Within the postural stability component of the VIS-REHAB protocol, there are static and dynamic balance exercises, along with general gross motor activities targeting core stability, agility, and bilateral coordination. The gaze stability part includes exercises enhancing oculomotor function such as smooth pursuit and saccadic movements, as well as VOR-exercises. Additionally, a general gross motor training program emphasises gaze stability by including exercises that improve eye-foot and eye-hand coordination. Furthermore, each session includes counselling and the provision of background information on the exercises.
  Arms: VIS-REHAB Protocol

SUMMARY:
The goal of this clinical trial is to investigate the short-term effect of a structured, combined postural control and gaze stabilisation protocol (VIS-REHAB protocol) in a group of vestibular-impaired children of different age categories (3-17 years). The main questions it aims to answer are:

* What is the short-term effect of the VIS-REHAB protocol?
* What are the most important factors that may influence the effect of and outcome after application of the VIS-REHAB protocol?

The participant will undergo both an active rehabilitation program (VIS-REHAB protocol) and a period during which physical therapy is discontinued (CTRL protocol).:

- VIS-REHAB protocol: Postural control (static and dynamic postural stability exercises), gaze stability exercises (oculomotor function and VOR-exercises) & general gross motor training with focus on gaze stability and postural control.

Researchers will compare the VIS-REHAB protocol with receiving no therapy (CTRL protocol) to evaluate potential enhancements in postural stability, gaze stability, motor performance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with identified vestibular dysfunction
* With or without concomitant hearing loss and/or cochlear implant (CI)

Exclusion Criteria:

* Children incapable to understand simple instructions (due to severe cognitive disorders, impaired language comprehension, etc.)
* Severe disorders of other primary sensory input systems for balance function
* Severe neuromotor disorders (incapable of independent standing and walking)
* Severe muscle tone disorders (e.g. cerebral palsy)
* Severe orthopaedic dysfunctions
* Patients with vision problems that cannot be corrected for
* Children with planned CI-surgery within 5 months before or during the study period

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Static postural stability and sensory integration as assessed by the Modified Clinical Test of Sensory Integration on Balance (mCTSIB) | Baseline and repeated before and after completing each 9-week protocol. There is a 1-week rest period between consecutive protocols.
  The child stands barefoot with feet together as still as possible for 30 seconds. There are eight test conditions: eyes open or closed, with or without foam, and eyes open or closed while on a foam, nodding the head in yaw or pitch at 0.33 Hz. The test will be conducted on a force platform, a Wii Balance Board (Nintendo Co., Ltd.), using the Colorado University BrainBLoX software. The total test time (s), anteroposterior and mediolateral sway (mm), centre of pressure path length (cm), sway velocity (m/s), and 95% confidence ellipse area (cm2 ) are measured by a custom-made code in MATLAB (The MathWorks, Inc. Natick, Massachusetts, United States).
Gaze stability as assessed by the Dynamic Visual Acuity (DVA) test | Baseline and repeated before and after completing each 9-week protocol. There is a 1-week rest period between consecutive protocols.
  The setup of the test is similar to that of the Static Visual Acuity (SVA) test, the only difference being that the patient's head will be passively moved by the examiner in the horizontal plane at a 2Hz-frequency over an amplitude of 15° from centre. The difference between the SVA and the DVA score will be included as output measure.

SECONDARY OUTCOMES:
Functional mobility and dynamic postural control during walking as assessed by the Timed Up and Go Test (TUG) | At the start of each 9-week protocol and at the very end of the complete trajectory (9-week protocol + 1-week rest period)
  Subjects sitting 3 m away from a 1m x 1m square with a cone in the centre, will be asked on the 'go' command to get up from the chair, walk to the square, navigate around the cone, come back to the chair and have a seat. Before the test, the procedure will be explained and demonstrated. Three trials will be conducted and the best time (recorded with stopwatch) will be used for analysis. Outcome parameters include the total test duration (s), number of steps, walking speed (m/s) and mean step length (cm).
Dynamic postural stability during walking as assessed by the Paediatric Modified Dynamic Gait Index (DGI) | At the start of each 9-week protocol and at the very end of the complete trajectory (9-week protocol + 1-week rest period)
  Subjects will be asked to complete 8 tasks, including walking on a flat surface, adjusting speed, and walking with horizontal and vertical head movements. It also evaluated walking over and around obstacles, turning while walking, and stepping on stairs. Each task is scored on a 3-point scale, with 3 indicating normal performance and 0 indicating severe impairment. The total score will serve as the outcome parameter.
Superior and inferior vestibular nerve and the functioning of the six semicircular canals, using the vestibulo-ocular reflex (VOR) assessed by the video Head Impulse Test (vHIT) | At the start of each 9-week protocol and at the very end of the complete trajectory (9-week protocol + 1-week rest period)
  The children will be instructed to sit on a chair and fixate an attractive visual target (i.e. movie on a tablet) at 1.50 m distance. Meanwhile the examiner will perform unpredictable head movements (10° - 20° amplitude) in, respectively, the horizontal, LARP (to stimulate the left anterior and right posterior canal), and RALP plane (to stimulate the right anterior and left posterior canal). Prior to interpretation of the results, the data will be thoroughly cleaned according to the following criteria: (1) head velocity between 120°/s (vertical) or 150°/s (horizontal) and 250°/s (upper limit for vertical and horizontal), and (2) head bounce below 25 % of the peak head velocity. The measured gain (of the VOR) (%), the symmetry between the left and right side (%), and the presence of covert/overt saccades (n, and % of the performed HITs) will be taken as outcome measures of this test.
Fine and gross motor skill assessment assessed by the Bruininks-Oseretsky Test of Motor Proficiency 2 (BOT-2) | At the start of each 9-week protocol and at the very end of the complete trajectory (9-week protocol + 1-week rest period)
  Each subtest yields an independent score, covering areas such as fine motor precision, fine motor integration, manual dexterity, upper-limb coordination, bilateral coordination, balance, running speed and agility, and strength. These individual scores contribute to composite scores for fine manual skills, manual coordination, body coordination, strength and agility, fine motor skills, gross motor skills, and overall motor performance, offering a comprehensive assessment of motor abilities.
Quality of life as assessed by the Paediatric Quality of Life Inventory (PedsQL) 4.0 | At the start of each 9-week protocol and at the very end of the complete trajectory (9-week protocol + 1-week rest period)
  . It is a 23-item inventory, applicable for (parents of) children from 2 to 18 year. It consists of four subdomains: (i) physical functioning (eight items), (ii) emotional functioning (five items), (iii) social functioning (five items), and (iv) school functioning (five items). Items are scored through a 5-point rating scale.
Static postural stability as assessed by the Single Leg Standing Test (SLS) | Baseline and repeated before and after completing each 9-week protocol. There is a 1-week rest period between consecutive protocols.
  Subjects will be instructed to stand on one leg as long as possible. After explanation and demonstration of the procedure, children will be granted one attempt (for 10 seconds) to get familiar with the exercise. SLS will be carried out both with eyes open and with eyes closed and three trials will be conducted. The test will be conducted on a force platform, a Wii Balance Board (Nintendo Co., Ltd.), using the Colorado University BrainBloX software. The total test time (s), anteroposterior and mediolateral sway (mm), centre of pressure path length (cm), sway velocity (m/s) and 95% confidence ellipse area (cm2).
Dynamic postural stability as assessed by the Paediatric Functional Reach Test | Baseline and repeated before and after completing each 9-week protocol. There is a 1-week rest period between consecutive protocols.
  After explanation and demonstration of the test, children will be granted one attempt to get familiar with the exercise. Children will be instructed to reach as far forward and sideward as possible with their hand(s) and without moving the feet. Three trials will be conducted in each condition. The furthest reaching point subtracted by the reaching distance in neutral, symmetrical posture will be included for analysis (cm).
Functional evaluation of the VOR by the Functional Head Impulse Test (fHIT) | Baseline and repeated before and after completing each 9-week protocol. There is a 1-week rest period between consecutive protocols.
  fHIT measurements will be conducted using the DVAstar Head Sensor (DIFRA Instrumentation, Eupen, Belgium) and accompanying software 'DiSoft II'. Participants will be seated 3 meters away from a visual target, and those who wear glasses or contact lenses will be encouraged to use them during the examination. The child must identify the orientation of the optotype (the letter 'C') that briefly appears on a computer screen for 80 milliseconds during unpredictable passive head movements (10 - 20° amplitude) in, respectively, the horizontal, LARP (to stimulate the left anterior and right posterior canal), and RALP plane (to stimulate the right anterior and left posterior canal). In each trial, the optotype is randomly rotated by 0°, 90°, 180°, or 270°. The size of the optotype corresponds to the SVA plus 0.6 LogMAR. The outcome parameter includes the percentage of correctly identified optotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Leen Maes, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Gent, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that will underlie the results reported in future publications of this study (text, tables, figures, and appendices) will be made available. The data will be available beginning 12 months and ending 36 months following the publication of the study results. Researchers who provide a methodologically sound proposal will be granted access. Proposals should be directed to marieke.fontaine@ugent.be. To gain access, data requestors will need to sign a data access agreement. The following documents will be available: study protocol, statistical analysis plan and informed consent forms. For further information or to submit a data access proposal, please contact marieke.fontaine@ugent.be.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 12 months and ending 36 months following the publication of study results.

REFERENCES:
- [Background] Melo RS, Lemos A, Paiva GS, Ithamar L, Lima MC, Eickmann SH, Ferraz KM, Belian RB. Vestibular rehabilitation exercises programs to improve the postural control, balance and gait of children with sensorineural hearing loss: A systematic review. Int J Pediatr Otorhinolaryngol. 2019 Dec;127:109650. doi: 10.1016/j.ijporl.2019.109650. Epub 2019 Aug 21. PMID 31466025
- [Background] Melo RS, Tavares-Netto AR, Delgado A, Wiesiolek CC, Ferraz KM, Belian RB. Does the practice of sports or recreational activities improve the balance and gait of children and adolescents with sensorineural hearing loss? A systematic review. Gait Posture. 2020 Mar;77:144-155. doi: 10.1016/j.gaitpost.2020.02.001. Epub 2020 Feb 3. PMID 32036319
- [Background] Melo RS, Lemos A, Delgado A, Raposo MCF, Ferraz KM, Belian RB. Use of Virtual Reality-Based Games to Improve Balance and Gait of Children and Adolescents with Sensorineural Hearing Loss: A Systematic Review and Meta-Analysis. Sensors (Basel). 2023 Jul 22;23(14):6601. doi: 10.3390/s23146601. PMID 37514897
- [Background] Martens S, Dhooge I, Dhondt C, Leyssens L, Sucaet M, Vanaudenaerde S, Rombaut L, Maes L. Vestibular Infant Screening - Flanders: The implementation of a standard vestibular screening protocol for hearing-impaired children in Flanders. Int J Pediatr Otorhinolaryngol. 2019 May;120:196-201. doi: 10.1016/j.ijporl.2019.02.033. Epub 2019 Feb 25. PMID 30849604
- [Derived] Fontaine M, Dhooge I, Dhondt C, Van Hecke R, Acke F, Van den Bossche L, Van Hoecke H, De Leenheer E, Maes L. Vestibular Infant Screening-Rehabilitation (VIS-REHAB): protocol for a randomised controlled trial on Vestibular Rehabilitation Therapy (VRT) in vestibular-impaired children. BMJ Open. 2024 Dec 20;14(12):e085575. doi: 10.1136/bmjopen-2024-085575. PMID 39806605